CLINICAL TRIAL: NCT06710236
Title: Evaluation of Investigational Hearing Instrument Features
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-26463
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Masking Description: Participants all receive the same intervention/hearing aid, but will be blinded as to which program they are being tested with.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Hearing Aid Users (Experimental): Participants will wear hearing instruments for the duration of the study period. They will be asked to complete questionnaires about their environment and experience.
  Interventions: Device: Hearing instrument

INTERVENTIONS:
Device: Hearing instrument — Conventional, daily wear hearing instruments will be used in this study.

SUMMARY:
The goal of this clinical trial is to learn how hearing instruments perform in varying environmental settings in adults with hearing loss. The main questions it aims to answer are:

How do varying versions of hearing instrument features perform based on exposure to different environments? What is the hearing instrument user preference between varying versions of hearing instrument features?

Participants will be fit with hearing instruments in the lab, and asked to wear them for the duration of the study period in their home environment. Participants will be asked to answer questionnaires throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 18 - 95 years
* N4 hearing loss
* Experienced hearing aid user
* English fluency
* Cognitively able to complete complex listening tasks

Exclusion Criteria:

* Normal hearing, or hearing loss outside the specified range
* No hearing aid experience
* Unable to speak, read, or write English fluently
* Cognitive impairment
* Any other condition or situation that impacts eligibility to participate in or complete study tasks, at the discretion of the investigator

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Hearing instrument feature performance | From enrollment to the completion of data collection, approximately 6 weeks
  Accuracy of hearing instrument feature performance based on environmental sampling and subjective reporting

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

IPD SHARING:
Plan to Share IPD: No